CLINICAL TRIAL: NCT04490512
Title: Randomised, Double-blind, Placebo-controlled Phase 1 Dose-escalation Study of FluBHPVE6E7 in HPV-16 Infected Women With Normal Cytology, CIN1 or CIN2
Brief Title: Study of FluBHPVE6E7 in HPV-16 Infected Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BlueSky Immunotherapies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BS-01
Record Dates: First submitted 2020-06-30; First posted 2020-07-29 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: HPV Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FluBHPVE6E7 (Experimental): Multiple administration of FluBHPVE6E7
  Interventions: Biological: FluBHPVE6E7
- Placebo (Placebo Comparator): Multiple administration of buffer solution
  Interventions: Biological: FluBHPVE6E7

INTERVENTIONS:
Biological: FluBHPVE6E7 — Multiple subcutaneous, intradermal or intramuscular administrations
  Other Names: Placebo

SUMMARY:
BS-01 is a randomised, double-blind, placebo-controlled, phase 1 dose escalation study assessing safety, tolerability and immunogenicity of FluBHPVE6E7, changes in the HPV infection status and cervical cytology, and biodistribution in HPV-16 infected women with normal cytology, CIN1 or CIN2. The safety and immunogenicity of two dose levels, 7.5 log10 and 9.0 log10 fTCID50/dose of FluBHPVE6E7 are assessed after three subcutaneous administrations. In addition the safety of 9.0 log10 fTCID50/dose of FluBHPVE6E7 is assessed after three intradermal or intramuscular administrations.

DETAILED DESCRIPTION:
BS-01 is a randomised, placebo-controlled, double- blind phase 1 dose-escalation study in women with normal cytology, CIN1 or CIN2.

The primary objective is to assess the safety and tolerability of FluBHPVE6E7. Secondary objectives are the assessment of the systemic immune responses to immunisations with FluBHPVE6E7, changes in HPV infection status and cervical cytology, and biodistribution.

Study medication is administered three times (Day 0, Week 4, Week 12). Study participants are randomised at a ratio of 3:1 for FluBHPVE6E7 or placebo. The first cohort is treated subcutaneously at dose level 7.5 log10 fTCID50/dose. The second cohort is treated subcutaneously at 9.0 log10 fTCID50/dose.

Interim safety reviews are performed by a Data Monitoring Committee. After completion of the dose-escalation and in order to collect additional safety data on the highest safe and tolerated dose level, additional study participants are enrolled into expansion cohorts treated three times subcutaneously, intradermally or intramuscularly at 9.0 log10 fTCID50/dose.

ELIGIBILITY:
Inclusion criteria:

* Females in general good health, EITHER 18-49 years of age with HPV-16 infection and cervical cytological evaluation with a normal result, OR 25-49 years of age, with HPV-16 infection, and histologically confirmed cervical intraepithelial neoplasia 1 (CIN1) or 2 (CIN2) for whom a "wait-and-see" approach for the study period is indicated
* HPV-16 infection has been confirmed at least twice by a validated HPV test separated by at least 3 months
* Satisfactory colposcopy (i.e. the entire cervix as well as the entire squamocolumnar junction can be visualized by colposcopy and there is no evidence of invasive cancer)
* No clinically significant out of range haematological, renal or hepatic laboratory tests
* Normal screening ECG or screening ECG with no clinically significant findings, as judged by the investigator
* Negative serum pregnancy test at screening
* Agree to use a reliable form of contraception during the whole study period. Reliable forms of contraception are hysterectomy or bilateral tubal ligation, hormonal methods (oral, injected, implanted or transdermal), intrauterine device, barrier method plus spermicide, history of a single male partner with vasectomy, or a history of abstinence deemed credible by the investigator. Furthermore, male partners should use condoms during the whole study period.
* Provides written informed consent

Exclusion criteria:

* Seropositivity (i.e. HAI titres >1:20) to the vector-derived wild type virus
* Any vaccination within 6 weeks of receiving study treatment
* Active significant viral infections including influenza, CMV, and EBV within 30 days of receiving study treatment
* Current cervical intraepithelial neoplasia 3 (CIN3)
* Co-infection with hepatitis B, hepatitis C, or HIV or having other immune deficient states
* Prior history of or current malignancy, high-grade cervical intraepithelial neoplasia (CIN2/3), vulvar intraepithelial neoplasia (VIN), vaginal intraepithelial neoplasia (VAIN), atypical glandular cells (AGC), adenocarcinoma in situ (AIS) or any suspicion of either micro-invasive or invasive disease
* Pregnancy, breastfeeding
* Influenza-like illness (ILI) during the preceding 3 months
* Known hypersensitivity to oseltamivir or any of its components
* Any anatomical condition of the cervix, including that resulting from previous cervical surgery, congenital malformation or other condition, that would interfere with a complete evaluation of the cervix
* Current pelvic inflammatory disease, cervicitis, or other gynaecological infection as per colposcopy and clinical examination
* Serious, concomitant disorder, including active systemic infection requiring treatment
* Presence of acute or chronic bleeding or clotting disorder, or use of blood thinners (e.g. anticoagulants or antiplatelet drugs) within 2 weeks of day 0
* A proven or suspected autoimmune disease
* Immunosuppression including any concurrent condition requiring the continued use of systemic or topical steroids, or the use of immunosuppressive agents, disease modifying doses of anti-rheumatic drugs (e.g., azathioprine, cyclophosphamide, cyclosporine, methotrexate), and biologic disease modifying drugs such as TNF-α inhibitors (e.g. infliximab, adalimumab or etanercept). Corticosteroids must be discontinued > 4 weeks prior to day 0 of study medication administration. Eye drops or ear drops containing corticosteroids are permissible.
* Acute or history of Herpes genitalis
* Prior major surgery within 4 weeks of day 0
* Administration of any blood product within 3 months of enrolment
* Any current significant cardiac, hepatic or renal disease or history of clinically significant, medically unstable disease (e.g. chronic renal failure; angina, myocardial ischemia or infarction, congestive heart failure, cardiomyopathy, or clinically significant arrhythmias)
* Any current or history of neurological disease including history of seizures
* Participation in another experimental protocol/use of investigational drug during the prior two months
* Any condition that, in the judgment of the investigator, might prevent safe participation in the study or interfere with study objectives
* Unability to comply with the protocol requirements

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (type, frequency, severity). | 7 days
  To assess the safety and tolerability of FluBHPVE6E7 by monitoring the type, frequency, and severity of AEs

SECONDARY OUTCOMES:
Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) following FluBHPVE6E7 administration | 16 weeks
  To evaluate of the induction of systemic vector-specific antibodies by HAI assay
Induction of HPV-specific T-cell response following FluBHPVE6E7 administration | 16 weeks
  To evaluate the induction of HPV16 E6- and E7-specific T-cells (%) by IFN-gamma ELISPOT analysis
Induction of HPV-specific CD4+ and CD8+ T-cells following FluBHPVE6E7 administration | 16 weeks
  To evaluate the induction of HPV16 E6- and E7 specific T-cells (%) by ICS and FACS analysis
Local HPV clearance | 16 weeks
  To evaluate the status of HPV-16 infection by HPV test (yes or no)
Cervical cytology | 16 weeks
  To evaluate changes in cervical cytology by Pap smear. Results are reported as Pap results according to the Bethesda System
Biodistribution: Detection of FluBHPVE6E7 in blood samples | 16 weeks
  To evaluate the presence of FluBHPVE6E7 by quantification of FluBHPVE6E7 genome copies in blood samples by RT-qPCR (copies per ml blood)
Biodistribution: Detection of FluBHPVE6E7 in nasal secretions | 16 weeks
  To evaluate the presence of FluBHPVE6E7 by qualitative real-time PCR assay specific for influenza B virus (positive or negative)
Number of participants with adverse events (type, frequency, severity). | 16 weeks
  To assess the safety and tolerability of FluBHPVE6E7 by monitoring the type, frequency, and severity of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria